CLINICAL TRIAL: NCT03306914
Title: Plasma Volume Expansion for Optimum Renal Transplant Surgery: Albumin Versus Starch
Brief Title: Comparing Human Albumin Versus Hydroxyethylstarch in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kareem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Albumin versus starch
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia Morbidity
MeSH Terms: interventions — zidovudine 5'-monophosphate-mannose-albumin conjugate; Albumins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin group (Active Comparator): Albumin resuscitation Albumin 5%
  Interventions: Other: Albumin resuscitation; Drug: Albumin 5%
- Hydroxyethylstarch group (Experimental): Hydroxyethylstarch resuscitation Hydroxyethylstarch 6%
  Interventions: Other: Hydroxyethylstarch resuscitation; Drug: Hydroxyethylstarch 6%

INTERVENTIONS:
Other: Albumin resuscitation — Albumin 5% is used as the intra-operative colloid
  Arms: Albumin group
Other: Hydroxyethylstarch resuscitation — Hydroxyethyl starch 6% is used as the intra-operative colloid
  Arms: Hydroxyethylstarch group
Drug: Albumin 5% — Infusion of Albumin 5% intra-operatively
  Other Names: Albumin
  Arms: Albumin group
Drug: Hydroxyethylstarch 6% — Infusion of Hydroxyethylstarch 6% intra-operatively
  Other Names: Tetraspan
  Arms: Hydroxyethylstarch group

SUMMARY:
In this study we try to review the possible effects when using modern hydroxyethylstarch solutions 6 % versus albumin 5% during living donor renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease, for living donor renal transplantation

Exclusion Criteria:

* severe cardiac or hepatic dysfunction, re-transplantation, coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of complications | 7 days
  Increased creatinine and/or need for dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kareem, Study Director — Kasr Al-Ainy Hospiral, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No